CLINICAL TRIAL: NCT05883618
Title: Global Neurotrauma Outcomes Study: Spine
Acronym: GNOS Spine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: NIHR Global Health Research Group on Neurotrauma (Unknown)
Responsible Party: Principal Investigator, Saniya Mediratta, Co-Principle Investigator, University of Cambridge
Other Study IDs: GNOSSpine
Record Dates: First submitted 2023-03-05; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Spine Injury; Trauma
Keywords: Traumatic spine injury; Global burden
MeSH Terms: conditions — Spinal Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiologically confirmed traumatic spine injury
  Interventions: Other: Exposure

INTERVENTIONS:
Other: Exposure — Human Development Index of Country

SUMMARY:
Primary aim:

Characterise case-mix, processes of care and variations in nonoperative and operative management strategies, including emergency, ward, surgical and ICU care, in patients presenting with traumatic spinal injury (TSI) between centres across low and high Human Development Index (HDI) countries.

Primary outcome measure:

The primary outcome measure will be Frankel Grade at 6 weeks post-admission (or discharge, whichever comes first).

Primary comparison:

Between country groups defined by human development index

Centre eligibility:

Any unit assessing patients with TSI worldwide will be eligible to participate

Patient eligibility:

All adult patients presenting with radiologically confirmed traumatic spinal injury.

Team:

Each participating unit will form a study team of up to four investigators including a study lead, local investigator 1/2 and an independent data validator.

Time period:

Local study teams may select any 30-day period from July 12th 2021 to start their study. Patients who meet the inclusion criteria between 00:01 on day 0 and 23:59 on day 30 of the selected study period will be included.

Validation:

There will be a two-phase data validation process. Phase 1 will be prospective, validating case ascertainment, and phase 2 will be retrospective, validating operative data.

DETAILED DESCRIPTION:
Background Traumatic spinal injury (TSI) accounts for a significant proportion of disability and death worldwide, with the majority of this burden affecting individuals in low- to middle- income countries. Crucially, to date, the current disease profile of TSI has not been characterised globally. In addition, the global approach to the care of patients following TSI is inconsistent with considerable geographical differences in process of care reported, and limited data available on the impact of these variations on outcomes following TSI. A better understanding of case-mix and processes of care is urgently needed to underpin efforts to identify ways of improving outcome relevant to different socioeconomic settings globally.

Objectives The primary objective of this study is to characterise the case-mix, processes of care and variations in nonoperative and operative management strategies, including emergency, ward, ICU care, in patients presenting with traumatic spinal injury (TSI) between centres across low and high Human Development Index (HDI) countries. The secondary aims are to summarise current local resources and management pathways for TSI through validation of provider profiling data, describe differences in indications for nonoperative and operative management, and short-term outcomes following TSI. This study aims to identify gaps in processes of care to identify targets for future interventions to improve TSI care across high and low-resource settings.

Methods A multi-centre, international, prospective, observational study. Any unit assessing patients with TSI worldwide will be eligible to participate. Each participating unit will form a study team responsible for gaining local approval, identifying patients for inclusion and conducting data collection. Data will be collected via a secure online platform in an anonymised form. Processes of care will be characterised by a detailed provider profiling exercise. A registry describing the case-mix and care of all adults presenting with radiologically confirmed TSI will be collected, in a given consecutive 30-day period during the study period starting in 2021.

Results The dataset, developed through an iterative feedback process involving clinicians from low and high Human Development Index (HDI) countries, includes patient demographics, details of injury mechanism, local injury management and, if applicable, timing and nature of surgery, post-operative care and immediate postoperative complications. Outcome measures include Frankel grade at 6 weeks post-admission (or at discharge or death, whichever event occurs first), early mortality, peri-operative complications, adverse events of special interest, functional status and mobility. Descriptive analyses of case-mix and the variations in processes of care will be conducted. Available resources, use of guidelines and variations in processes of care will be characterised using both provider profiling responses and patient-level data collected. Areas where known best practice is deficient or unavailable will be identified as potential targets for future implementation studies.

Conclusions GNOS Spine aims to provide a global snapshot of the case-mix, management, processes of care and short-term outcomes of patients presenting with TSI. In addition, the study aims to identify areas for further study, and establish a platform and clinical network to facilitate this future research in global neurotrauma and spinal surgery.

ELIGIBILITY:
Centre inclusion Criteria

* Any primary, secondary or tertiary institution worldwide managing patients with TSI is eligible to participate.
* In many institutions, management for TSI may be provided by spinal surgeons - however, centres in which management for TSI is provided by general surgeons, trauma surgeons, general medical doctors or even non-physician clinicians are also eligible to participate.

Patient inclusion and exclusion criteria Inclusion Criteria

* All adult patients presenting to the participating institution with a first presentation of TSI confirmed radiographically, during the selected 30-day inclusion period are eligible for inclusion in the core study.

Exclusion Criteria

* Elective (planned) or semi-elective (patient initially discharged after emergency with planned
* intervention at a future date) admissions
* Patients who have previously had an admission for TSI rendering them eligible for inclusion in this study (regardless of whether they were included on the previous admission or not)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with radiologically confirmed traumatic spine injury
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Frankel Grade | At discharge or 6 weeks post-admission, whichever comes first
  A = complete motor and sensory loss (poor outcome), E = no neurological symptoms or signs (good outcome)

SECONDARY OUTCOMES:
Mortality | At discharge or 6 weeks post-admission, whichever comes first
  Assessment of survival
Length of Stay | At discharge or at 6 weeks post-admission (whichever comes first)
  Hospital and ICU
Peri-operative Complications | At discharge or at 6 weeks post-admission (whichever comes first)
  Return to operating theatre, surgical site infections, adverse events of special interest (pressure ulcer, pneumonia, DVT)
Independence with activities of daily living (ADLs) | At discharge or at 6 weeks post-admission (whichever comes first)
  Rating of specific ADLs as unaided, with aid or completely dependent
Mobility | At discharge or at 6 weeks post-admission (whichever comes first)
  Mechanism of mobility e.g. mobilising independently, mobilising with a frame, wheelchair, bed bound etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Saniya Mediratta, Principal Investigator — NIHR Global Health Research Group on Neurotrauma; Jibin Francis, Principal Investigator — NIHR Global Health Research Group on Neurotrauma; Peter Hutchinson, Principal Investigator — NIHR Global Health Research Group on Neurotrauma; Rikin Trivedi, Principal Investigator — NIHR Global Health Research Group on Neurotrauma
Locations (1):
- University of Cambridge, Cambridge, County, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After publication of the main results, the pooled dataset will be available to all members of the GNOS Spine collaboration for secondary analysis, after judgement and approval of each proposed analysis by the central study team.
Supporting Information: Study Protocol, SAP
Time Frame: Following publication of the main results

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT05883618/Prot_SAP_000.pdf